CLINICAL TRIAL: NCT01618487
Title: Comparison of Surgical Interventions for Lateral Epicondylitis: A Randomized, Prospective Study
Brief Title: Comparison of Surgical Interventions for Lateral Epicondylitis: A Prospective Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Christine M. Kleinert Institute for Hand and Microsurgery (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11.0565
Record Dates: First submitted 2012-06-11; First posted 2012-06-13 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Lateral Epicondylitis; Tennis Elbow
Keywords: tennis elbow; lateral epicondylitis
MeSH Terms: conditions — Tennis Elbow | interventions — Debridement; Wound Healing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arthroscopic tenotomy (Active Comparator): Patients who are in this group will have arthroscopic tenotomy. A scope is used to see the tendon and release it.
  Interventions: Procedure: Arthroscopic tenotomy
- Open tenotomy (Active Comparator): Patients in this group will undergo open tenotomy. This involves opening the skin to expose the muscle and tendon, and then the tendon is released.
  Interventions: Procedure: Open tenotomy
- Debridement and repair (Active Comparator): The patients in this group will undergo an arthroscopic technique (scope and small incision) to go in and remove any tissue that is diseased/does not belong and repair the tear(s) in the tendon.
  Interventions: Procedure: Debridement and repair

INTERVENTIONS:
Procedure: Arthroscopic tenotomy — This is a surgical procedure where small incisions are made and a scope is used to see the tendon and release it.
  Arms: Arthroscopic tenotomy
Procedure: Open tenotomy — This involves opening the skin on the arm up to expose the muscle and tendon. There is a total of 1 incision made.
  Arms: Open tenotomy
Procedure: Debridement and repair — This involves using an arthroscopic technique (using a scope and a small incision) to go in and remove any tissue that is diseased/does not belong and repairing the tear(s) in the tendon. There is a total of 1-2 incisions made.
  Arms: Debridement and repair

SUMMARY:
The investigator hopes to determine if one of three current standard of care surgeries for lateral epicondylitis (tennis elbow) is more effective than others. The three surgeries are: arthroscopic tenotomy, open tenotomy, and debridement and repair.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 yrs old
* pain over the lateral epicondyle (via palpitation over the lateral epicondyle, resisted wrist extension, resisted finger extension of the middle finger) for a duration of greater than 6 months prior to enrollment
* conservative treatment has failed and surgical intervention is recommend as standard of care
* ability to give informed consent

Exclusion Criteria:

* had surgery by a physician or specialist within the last 2 years as treatment for lateral epicondylitis
* congenital deformities, tendon ruptures or elbow fractures within the past year
* co-existing elbow diagnosis (i.e. osteoarthritis or instability)
* pregnant women, women trying to get pregnant, or breastfeeding mothers
* under the age of 18 or over 65
* incapable of giving informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2012-02; Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
symptom severity and functional outcome score (Patient Rated Tennis Elbow Evaluation) | 24 months
  The primary outcome measure will be the difference btetwee the pre and post operative assessments of questionnaire and symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: Tuna Ozyurekoglu, MD, Principal Investigator — Christine M. Kleinert Institute of Hand and Microsurgery
Locations (1):
- Christine M. Kleinert Institute of Hand and Microsurgery, Louisville, Kentucky, United States